CLINICAL TRIAL: NCT04636268
Title: A Prospective, Multicenter, Open-label, Single-arm Study to Evaluate the Efficacy and Safety of Human Plasma-derived Fibrinogen Concentrate (FIB Grifols) in Subjects With Congenital Afibrinogenaemia and Severe Hypofibrinogenemia Requiring Either On-demand Treatment for Acute Bleeding or Surgical Prophylaxis
Brief Title: FIB Grifols Congenital Deficiency for On-demand Treatment and Surgical Prophylaxis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to a business decision.
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Therapeutics LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC1801; 2018-004005-81 (EudraCT Number)
Record Dates: First submitted 2020-03-16; First posted 2020-11-19 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Congenital Afibrinogenemia; Hypofibrinogenemia
MeSH Terms: conditions — Afibrinogenemia | interventions — Fibrinogen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FIB Grifols (Experimental): FIB Grifols is the IP and will be administered via slow intravenous (IV) infusion at a rate not to exceed 5 mL/minute.
  Dosing will be individually calculated for each subject based on the target plasma fibrinogen level according to the type of bleeding, measured actual plasma fibrinogen level before infusion, and body weight. The IP will be administered according to the nominal potency of the product.
  Interventions: Biological: FIB Grifols

INTERVENTIONS:
Biological: FIB Grifols — FIB Grifols is the IP and will be administered via slow intravenous (IV) infusion at a rate not to exceed 5 mL/minute.
  Dosing will be individually calculated for each subject based on the target plasma fibrinogen level according to the type of bleeding, measured actual plasma fibrinogen level before infusion, and body weight. The IP will be administered according to the nominal potency of the product.
  Other Names: Fibrinogen

SUMMARY:
This is a phase 3, multi-center, prospective, open-label, single-arm, clinical trial to be carried out in subjects with congenital fibrinogen deficiency manifested as afibrinogenemia or severe hypofibrinogenemia.

This clinical trial is planned to be performed at study sites in multiple countries. It is planned to include a maximum of 32 adult and pediatric subjects with congenital fibrinogen deficiency in order to provide at least 28 evaluable acute bleeding episodes and/or surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject between 6 to 70 years of age.
2. Signed and dated written ICF, or the subject's parent or legal guardian signs and dates the ICF where applicable, and the Subject Authorization Form (SAF) where applicable. Pediatric subjects, as defined by local regulations, will be asked to sign an age appropriate assent form.
3. Diagnosed with congenital fibrinogen deficiency manifested as afibrinogenemia or severe hypofibrinogenemia (fibrinogen <50 mg/dL) and expected to require treatment for acute bleeding (either spontaneous or after trauma [defined as any accidental event leading to acute bleeding]), or prophylaxis of bleeding before a surgical intervention or invasive procedure.
4. Fibrinogen level < 50 mg/dL determined by Clauss method at baseline (sample drawn within 24 hours prior to infusion on Infusion 1 Day 1 Visit).
5. Female subjects of child-bearing potential must have a negative test for pregnancy blood or urine human chorionic gonadotropin (HCG)-based assay at baseline (sample drawn within 24 hours prior to infusion on Infusion 1 Day 1 Visit).
6. Willing to comply with all aspects of the clinical trial protocol, including blood sampling, for the entire duration of the study.

Exclusion Criteria:

1. Has acquired (secondary) fibrinogen deficiency.
2. Diagnosed with dysfibrinogenemia.
3. Has known antibodies against fibrinogen.
4. Has history of anaphylaxis or severe systemic response to any drug or blood-derived product.
5. Has history of intolerance to any component of the IP.
6. Documented history of immunoglobulin A (IgA) deficiency and antibodies against IgA.
7. Is a female who is pregnant, breastfeeding or, if of child-bearing potential, unwilling to practice a highly effective method of contraception (eg, oral, injectable, or implantable hormonal methods of contraception, placement of an IUD or intrauterine system, condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization, or true abstinancea) throughout the study.
8. Has any medical condition which is likely to interfere with the evaluation of the IP and/or the satisfactory conduct of the clinical trial according to the investigator's judgment.
9. Has congenital or acquired bleeding disorders other than congenital fibrinogen deficiency.
10. Has life expectancy of less than 6 months.
11. Received FRT within 21 days prior to the Screening Visit.
12. Receiving, or having received within 3 months prior to the Screening Visit of this clinical trial, any investigational drug or device.
13. Is unlikely to adhere the protocol requirements, or is likely to be uncooperative, or unable to provide a storage sample prior to IP infusion.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Hemostatic efficacy of FIB Grifols in on-demand treatment of all documented acute bleeding episodes as assessed by the Independent Endpoint Adjudication Committee (IEAC) Using a 4-Point Scale | Up to Day 7
  To clinically evaluate the hemostatic efficacy of FIB Grifols in on-demand treatment of all documented acute bleeding episodes in subjects with congenital fibrinogen deficiency as determined by the the proportion of successful treatment responses (Yes/No) indicated by a hemostatic efficacy rating of "Excellent" or "Good" as assessed by the IEAC using a 4 point scale. Hemostatic efficacy will be determined at end of treatment observation period (either at Day 3 for non-life threatening bleeding episodes, at Day 7 for life-threatening bleeding episodes, or at 24 hours after the end of the last infusion of FIB Grifols, whichever is later).
Hemostatic efficacy of FIB Grifols in perioperative management of bleeding during and after all documented surgical procedures as assessed by the IEAC Using a 4-Point Scale | Up to Day 7
  To clinically evaluate the hemostatic efficacy of FIB Grifols in the perioperative management of bleeding during and after all documented surgical procedures in subjects with congenital fibrinogen deficiency as determined by the the proportion of successful treatment responses (Yes/No) indicate by an adjudicated hemostatic efficacy rating of "Success" in preventing excessive bleeding during and after all documented surgical procedures as assessed by the IEAC using a 4 point scale. Hemostatic efficacy will be determined at end of treatment observation period (either at Day 3 for minor surgical procedures, at Day 7 for major surgical procedures, or at 24 hours after the end of the last infusion of FIB Grifols, whichever is later).

SECONDARY OUTCOMES:
Hemostatic Efficacy of FIB Grifols in Treating the First Documented Acute Bleeding Episode as Assessed by the IEAC Using a 4-Point Scale. | Up to Day 7
  Overall clinical assessment of the hemostatic efficacy of FIB Grifols in treating the first documented acute bleeding episode using a 4-point hemostatic efficacy scale including the four items: 'excellent,' 'good,' moderate,' and 'none'. These data will be transformed into a dichotomous result, with 'treatment success-yes' defined as a rating of 'excellent' or 'good' and 'treatment success-no' defined as a rating of 'moderate' or 'none'. This secondary efficacy endpoint will be assessed by the IEAC.
  Hemostatic efficacy will be determined at end of treatment observation period (either at Day 3 for non-life threatening bleeding episodes, at Day 7 for life-threatening bleeding episodes, or at 24 hours after the end of the last infusion of FIB Grifols, whichever is later).
Hemostatic Efficacy of FIB Grifols in Preventing Excessive Bleeding During and After the First Documented Surgical Procedure as Assessed by the IEAC Using a 4-Point Scale | Up to Day 7
  Overall clinical assessment of the hemostatic efficacy of FIB Grifols in preventing excessive bleeding during and after the first documented surgical procedure using a 4-point hemostatic efficacy scale including the four items: 'excellent,' 'good,' moderate,' and 'none'. These data will be transformed into a dichotomous result, with 'treatment success-yes' defined as a rating of 'excellent' or 'good' and 'treatment success-no' defined as a rating of 'moderate' or 'none'. This secondary efficacy endpoint will be assessed by the IEAC.
  Hemostatic efficacy will be determined at end of treatment observation period (either at Day 3 for minor surgical procedures, at Day 7 for major surgical procedures, or at 24 hours after the end of the last infusion of FIB Grifols, whichever is later).
Hemostatic Efficacy of FIB Grifols in Treating the First Acute Bleeding Episode | Up to Day 7
  Overall clinical assessment of the hemostatic efficacy of FIB Grifols in treating the first acute bleeding episode as assessed by the principal investigator at each trial site using a 4-point hemostatic efficacy scale including the four items: 'excellent,' 'good,' moderate,' and 'none'. These data will be transformed into a dichotomous result, with 'treatment success-yes' defined as a rating of 'excellent' or 'good' and 'treatment success-no' defined as a rating of 'moderate' or 'none'.
  Hemostatic efficacy will be determined at end of treatment observation period (either at Day 3 for non-life threatening bleeding episodes, at Day 7 for life-threatening bleeding episodes, or at 24 hours after the end of the last infusion of FIB Grifols, whichever is later).
Hemostatic Efficacy of FIB Grifols in Treating All Acute Bleeding Episodes | Up to Day 7
  Overall clinical assessment of the hemostatic efficacy of FIB Grifols in treating all acute bleeding episodes as assessed by the principal investigator at each trial site using a 4-point hemostatic efficacy scale including the four items: 'excellent,' 'good,' moderate,' and 'none'. These data will be transformed into a dichotomous result, with 'treatment success-yes' defined as a rating of 'excellent' or 'good' and 'treatment success-no' defined as a rating of 'moderate' or 'none'.
  Hemostatic efficacy will be determined at end of treatment observation period (either at Day 3 for non-life threatening bleeding episodes, at Day 7 for life-threatening bleeding episodes, or at 24 hours after the end of the last infusion of FIB Grifols, whichever is later).
Hemostatic Efficacy of FIB Grifols in Preventing Excessive Bleeding Intra-operatively for All Surgical Procedures. | Up to Day 7
  Clinical assessment of the hemostatic efficacy of FIB Grifols in preventing excessive bleeding intra-operatively for all surgical procedures as assessed by the surgeon (defined as the licensed medical professional performing the invasive procedure [eg, dentist]) using a 4-point hemostatic efficacy scale including the four items: 'excellent,' 'good,' moderate,' and 'none'. These data will be transformed into a dichotomous result, with 'treatment success-yes' defined as a rating of 'excellent' or 'good' and 'treatment success-no' defined as a rating of 'moderate' or 'none'.
  Hemostatic efficacy will be determined at end of treatment observation period (either at Day 3 for minor surgical procedures, at Day 7 for major surgical procedures, or at 24 hours after the end of the last infusion of FIB Grifols, whichever is later).
Hemostatic Efficacy of FIB Grifols in Preventing Excessive Bleeding After All Surgical Procedures (ie, Post-operative) | Up to Day 7
  Clinical assessment of the hemostatic efficacy of FIB Grifols in preventing excessive bleeding after all surgical procedures (ie, post-operative) as assessed by the principal investigator at each trial site using a 4-point hemostatic efficacy scale including the four items: 'excellent,' 'good,' moderate,' and 'none'. These data will be transformed into a dichotomous result, with 'treatment success-yes' defined as a rating of 'excellent' or 'good' and 'treatment success-no' defined as a rating of 'moderate' or 'none'.
  Hemostatic efficacy will be determined at end of treatment observation period (either at Day 3 for minor surgical procedures, at Day 7 for major surgical procedures, or at 24 hours after the end of the last infusion of FIB Grifols, whichever is later).